CLINICAL TRIAL: NCT03728504
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of ASN002 in Subjects With Moderate To Severe Chronic Hand Eczema Refractory to Corticosteroid Therapy
Brief Title: Study to Evaluate ASN002 in Subjects With Moderate To Severe Chronic Hand Eczema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asana BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASN002AD-202
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Chronic Hand Dermatitis
Keywords: eczema; hand eczema; hand dermatitis
MeSH Terms: conditions — Eczema | interventions — gusacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ASN002 40 mg (Experimental): 40 mg ASN002
  Interventions: Drug: ASN002
- ASN002 80 mg (Experimental): 80 mg ASN002
  Interventions: Drug: ASN002
- Placebo oral tablet (Placebo Comparator): Matching placebo for ASN002 doses
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: ASN002 — Daily dose of ASN002 for 32 weeks
  Arms: ASN002 40 mg; ASN002 80 mg
Drug: Placebo Oral Tablet — Daily dose of Placebo Oral Tablet for 16 weeks
  Arms: Placebo oral tablet

SUMMARY:
Randomized double-blind/placebo study to evaluate the efficacy of ASN002 in subjects with severe chronic hand eczema.

DETAILED DESCRIPTION:
This is a placebo controlled study where subjects with severe chronic hand eczema will be randomized (1:1:1) to receive ASN002 at 40 mg, 80 mg, or placebo once daily for 16 weeks (Part A). Then, in Part B, subjects who were assigned to placebo in the first part of the study will receive the highest dose of ASN002 (80 mg) for the rest of the treatment period (up to Week 32). The subjects who were assigned ASN002 in the first part of the study will continue on the same assigned treatment dose during the second part of the study (Week 16 to Week 32). The total treatment period of 32 weeks will be followed by a 4 week follow-up period.This study will also characterize the pharmacokinetics and pharmacodynamics of ASN002 through blood sampling and three or four biopsies from subjects who consent.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any study-related procedure being performed
* Male or female subject, aged 18 to 75 years, inclusive, at the time of consent.
* Subject has a history of severe CHE for at least 6 months prior to baseline
* Subject has hand eczema refractory to high potency or ultra-high potency topical corticosteroids
* Subject has moderate to severe CHE at Day 1, as defined by a hand PGA 3 or 4.
* Subject has been using an emollient on their hands and feet (except those containing urea or salicylic acid) every day at the same frequency for at least 1 week prior to Day 1
* Subject has a body mass index (BMI) ≤ 38 kg/m2.
* Female subject of childbearing potential has had a negative serum pregnancy test at screening and negative urine pregnancy test on Day 1.
* Willing and able to comply with clinical visits and study related procedures.

Exclusion Criteria:

* Presence of any of the following laboratory abnormalities at the screening visit: Hemoglobin < 11 g/dL, White blood cell (WBC) < 3.0 x 103 /μL, Platelet count < 125 x 103 /μL, Neutrophils < 1.80 x 103 /μL, Lymphocytes <0.9 x 103 /μL, Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2x the upper limit of normal (ULN),Total bilirubin > 1.2x ULN (except for elevated indirect bilirubin secondary to Gilbert's syndrome), Creatinine > ULN
* A serious uncontrolled condition including hypertension, active tuberculosis, hepatitis B or C infection, immune deficiency, heart disease, heart conduction disorder, diverticulitis, diabetes, reflux disease requiring protocol pump inhibitor therapy, malabsorption syndrome, or cancer.
* Active skin infections of the hands and/or feet
* Any medical or psychiatric condition which, in the opinion of the investigator or the sponsor's medical monitor, would place the patient at risk, interfere with participation in the study, or interfere with the interpretation of study results
* Pregnant or breast-feeding women
* Known hypersensitivity to ASN002 or its excipients
* Prior treatment with SYK or JAK inhibitors for which the subject received no clinical benefit, or the subject relapsed whilst on therapy.
* Subject has received any marketed or investigational biological agent within 12 weeks or 5 half-lives (whichever is longer) prior to Day 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Zammit, Ph.D., Study Director — Asana BioSciences
Locations (23):
- United States (17):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Dermatology Research Associates, Los Angeles, California
  - Sweet Hope Research Specialty, Inc, Hialeah, Florida
  - RM Medical Research, Inc., Miami, Florida
  - Advanced Clinical Research, Boise, Idaho
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - Dermatology Specialists Research, Louisville, Kentucky
  - DelRicht Research, New Orleans, Louisiana
  - Maryland Laser Skin and Vein, Hunt Valley, Maryland
  - BTC Network, Fort Gratiot, Michigan
  - Minnesota Clinical Research Center, Fridley, Minnesota
  - ActivMed Practices and Research, Inc., Portsmouth, New Hampshire
  - Dermatologists of Greater Colombus, Bexley, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Progressive Clinical Research, San Antonio, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Dermatology Specialists of Spokane, Spokane, Washington
- Canada (6):
  - SimcoDerm Medical and Surgical Dermatology Centre, Barrie, Ontario
  - Wei Jing Loo Medicine Professional Corp., London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - G. Daniel Schachter Medicine Professional, Toronto, Ontario
  - Innovaderm Research, Inc., Montreal
  - Centre de Recherche Dermatologique du Quebec metropolitain, Québec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bar J, Del Duca E, David E, Bose S, Chefitz G, Brunner PM, Bissonnette R, Guttman-Yassky E. Skin Tape Stripping Reveals Distinct Biomarker Profiles in Chronic Hand Eczema of Patients With and Without Comorbid Atopic Dermatitis. Allergy. 2025 Aug;80(8):2271-2285. doi: 10.1111/all.16466. Epub 2025 Jan 6. PMID 39760239

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ASN002 40 mg | ASN002 80 mg | Placebo Oral Tablet
Started | 33 | 32 | 32
Completed | 27 | 19 | 22
Not Completed | 6 | 13 | 10

BASELINE CHARACTERISTICS:
Groups:
- ASN002 40 mg: 40 mg ASN002
  ASN002: Daily dose of ASN002
- ASN002 80 mg: 80 mg ASN002
  ASN002: Daily dose of ASN002
- Placebo Oral Tablet: Matching placebo for ASN002 doses
  Placebo Oral Tablet: Daily dose of Placebo
- Total: Total of all reporting groups
Arm/Group | ASN002 40 mg | ASN002 80 mg | Placebo Oral Tablet | Total
Number analyzed (Participants) | 33 | 32 | 32 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 29 | 83
  >=65 years | 6 | 5 | 3 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (16.86) | 46.7 (15.76) | 41.8 (16.64) | 44.2 (16.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 18 | 65
  Male | 10 | 8 | 14 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 2 | 13
  Not Hispanic or Latino | 30 | 24 | 30 | 84
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 2 | 9
  White | 27 | 27 | 28 | 82
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 11 | 10 | 29
  United States | 25 | 21 | 22 | 68
modified Total Lesion Symptom Score (mTLSS) [Mean (Standard Deviation); unit: units on a scale] — The modified total lesion symptom score (mTLSS) is an assessment of the severity of each of the following: erythema, scaling, lichenification/hyperkeratosis, vesicles, edema, fissures, and pruritus/pain. Each of these are rated using a 4-point severity scale. The ratings are added to create a total mTLSS calculated as the sum of assigned individual scores with a maximum value of 21 (most severe disease) and a minimum of 0 (no disease)
  units on a scale | 13.2 (3.42) | 13.5 (2.57) | 13.0 (3.41) | 13.2 (3.13)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Modified Total Lesion Symptom Score (mTLSS)
Description: Percent change from baseline in hand mTLSS at Week 16. The mTLSS is an assessment of the severity of each of the following: erythema, scaling, lichenification/hyperkeratosis, vesicles, edema, fissures, and pruritus/pain. Each of these are rated using a 4-point severity scale. The ratings are added to create a total mTLSS calculated as the sum of assigned individual scores with a maximum value of 21 (most severe disease) and a minimum of 0 (no disease)
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | ASN002 40 mg | ASN002 80 mg | Placebo Oral Tablet
Number analyzed (Participants) | 33 | 32 | 32
percentage change | -49.5 (40.65) | -71.3 (26.97) | -29.9 (38.51)

2. Secondary Outcome: Change From Baseline in Hand Physician Global Assessment (PGA)
Description: Proportion of participants with a response of Physicians Global Assessment achieving clear (0) or almost clear (1)
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ASN002 40 mg | ASN002 80 mg | Placebo Oral Tablet
Number analyzed (Participants) | 33 | 32 | 32
Participants | 7 | 10 | 2

3. Secondary Outcome: Change From Baseline in Hand Patient Global Assessment (PaGA)
Description: Reduction of PaGA compared to baseline where marked improvement was noted with at least 75% clear
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ASN002 40 mg | ASN002 80 mg | Placebo Oral Tablet
Number analyzed (Participants) | 33 | 32 | 32
Participants | 7 | 7 | 2

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | ASN002 40 mg | ASN002 80 mg | Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/33 | 2/32 | 1/32
Other Adverse Events (participants affected / at risk) | 19/33 | 24/32 | 17/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ASN002 40 mg (N=33) | ASN002 80 mg (N=32) | Placebo Oral Tablet (N=32)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alcoholism (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ASN002 40 mg (N=33) | ASN002 80 mg (N=32) | Placebo Oral Tablet (N=32)
Upper respiratory tract infection (Infections and infestations) | 5 | 2 | 3
Nasopharyngitis (Infections and infestations) | 2 | 3 | 2
Headache (Nervous system disorders) | 5 | 6 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0
Hypersensitivity (Immune system disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Ear Infection (Infections and infestations) | 0 | 1 | 0
Eyelid infection (Infections and infestations) | 0 | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pilonidal cyst (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Granuloma annulare (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash generalized (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 1
Peripheral swelling (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 2 | 0
Face oedema (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Thirst (General disorders) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood CPK increased (Investigations) | 1 | 1 | 0
Blood potassium increased (Investigations) | 2 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 0
Reticulocyte count decreased (Investigations) | 0 | 1 | 0
Weight increased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Wisdom teeth removal (Surgical and medical procedures) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT03728504/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/04/NCT03728504/SAP_001.pdf